CLINICAL TRIAL: NCT05261763
Title: Study on the Effects of Trigger Point Dry Needling on Patients With Patello-femoral Pain Syndrome: A Randomized Controlled Trial
Brief Title: Effects of Trigger Point Dry Needling in Individuals With Patello Femoral Pain Syndrome : A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC-FSD-00238
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Patellofemoral Pain Syndrome; Dry Needling; Trigger Points
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A will receive trigger point dry needling in quadricep muscles
  Interventions: Other: Dry Needling
- Group B (Sham Comparator): Group B will get Sham needling in quadriceps muscles
  Interventions: Other: Sham Dry Needing

INTERVENTIONS:
Other: Dry Needling — abc
  Arms: Group A
Other: Sham Dry Needing — xyz
  Arms: Group B

SUMMARY:
A double blinded clinical controlled trial will be performed on individuals with patello femoral pain syndrome in which Trigger Point Dry Needling will be given to experimental group while Sham Needling will be given to the control group, targeting the trigger points present in the Quadriceps of affected individuals assessing the pain,functional disability and range of motion of the affected individuals.

DETAILED DESCRIPTION:
A double blinded Randomized Controlled Trial of 6 months study after the approval of synopsis, will be conducted. Convenience sampling technique will be used to enroll the patients. Patients will be selected according to predefined inclusion and exclusion criteria. All patients who fulfill inclusion criteria will be allocated in two group through randomization by lottery method. Group A will receive TrP-DN and group B will receive Sham Needling. Both groups will be asked to perform stretching exercise of Quadriceps daily after needling. The patients' outcomes will be measured by VAS for pain intensity and Kujala Questionnaire for functional status. The comparison between pre-treatment and post-treatment data will be done after 3 months. Informed consents will be taken from each patient. Data entry and analysis will be done with SPSS 23.

ELIGIBILITY:
Inclusion Criteria:

- 1. Both genders 2. Ages range from 18-40 years 3. They have clinical diagnosis of PFPS (the diagnosis was confirmed by a positive patellar grind test and tenderness of medial and lateral patellar facets) 4. Participants are also required to have a minimum pain score of 3 on Numeric Pain Scale 5. Kujala patellofemoral questionnaire score of 50 to 80 before the intervention.

6. Patients willing to participate

Exclusion Criteria:

* History of any following conditions

  1. Participants who have received any treatment for PFPS within the 3 months
  2. A history of lower extremities fracture or surgery
  3. Presence of MSK diseases such as Acute Herniated Disc or Spondylolisthesis
  4. History of any chronic disease e.g. Diabetes Mellitus

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 8th week
  Visual Analogue Scale
Kujala Questionnaire | 8th week
  functional disability will be check by Kujala Questionnaire
Goniometer | 8th week
  range of motion will be checked by Goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neal BS, Lack SD, Lankhorst NE, Raye A, Morrissey D, van Middelkoop M. Risk factors for patellofemoral pain: a systematic review and meta-analysis. Br J Sports Med. 2019 Mar;53(5):270-281. doi: 10.1136/bjsports-2017-098890. Epub 2018 Sep 21. PMID 30242107
- [Background] Erratum: Effects of Trigger Point Dry Needling on Neuromuscular Performance and Pain of Individuals Affected by Patellofemoral Pain: A Randomized Controlled Trial [Corrigendum]. J Pain Res. 2020 Sep 7;13:2237. doi: 10.2147/JPR.S278493. eCollection 2020. PMID 32982385
- [Background] Mason JS, Crowell M, Dolbeer J, Morris J, Terry A, Koppenhaver S, Goss DL. THE EFFECTIVENESS OF DRY NEEDLING AND STRETCHING VS. STRETCHING ALONE ON HAMSTRING FLEXIBILITY IN PATIENTS WITH KNEE PAIN: A RANDOMIZED CONTROLLED TRIAL. Int J Sports Phys Ther. 2016 Oct;11(5):672-683. PMID 27757280